CLINICAL TRIAL: NCT00190229
Title: CESAR (Randomized Therapeutic Study of Steroid vs. Steroid Plus Cyclosphosphamide for Severe Viscera Henoch-Schoenlein Purpura)
Brief Title: Efficacy of Steroid Versus Steroid Plus Cyclophosphamide for Severe Henoch-Schoenlein Purpura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel OUSLIMANI, Department Clinical Research of developpement
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P011014
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2007-03

CONDITIONS: Henoch-Schoenlein Purpura
Keywords: Vasculitis; Cyclophosphamide; Renal failure
MeSH Terms: conditions — IgA Vasculitis; Vasculitis; Renal Insufficiency | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide

SUMMARY:
Henoch-Schonlein purpura is a leucocytoclastic systemic vasculitis involving small vessels with the deposition of immune complexes containing IgA. It is characterized by the association of skin, joint and gastrointestinal manifestations. Even though the evolution is usually simple, some patients, especially adults, may have severe visceral involvement including heart, lung, brain and renal disease. The best treatment is currently unknown. This study will test the safety and efficacy of steroids associated or not with cyclosphosphamide to treat the acute lesions and to prevent the development of chronic lesions.

DETAILED DESCRIPTION:
The protocol test the role of 2 modalities of treatment (steroid vs. steroid and cyclophosphamide) for severe systemic form of Henoch-Schonlein purpura. The severe forms include extracapillary glomerulonephritis, myocarditis, pneumonitis, occult involvement, severe gastro-intestinal bleeding. No other randomized trial has been performed in adult patient for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Henoch-Schoenlein purpura
* Patient's age > 18 years

Exclusion criteria:

* Patient presenting a purpura RHEUMATOID the diagnosis of which is confirmed by the histology presenting at least a visceral infringement(achievement) making consider the affection as engraves(burns)
* of 18 or more years old Patient
* Patient capable of understanding(including) the advantages and the risks of the try
* Patient having given his assent lit in writing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Birmingham Vasculitis Activity Score (BVAS) | during de study
  Birmingham Vasculitis Activity Score (BVAS)

SECONDARY OUTCOMES:
Chronic lesions (Vasculitis Damage Index) | during the study
  Chronic lesions (Vasculitis Damage Index)
Renal function at 12 months | during the study
  Renal function at 12 months
Kidney survival at 12 months | during the study
  Kidney survival at 12 months
Patient survival at 12 months | during the study
  Patient survival at 12 months
Blood pressure | during th study
  Blood pressure
Infections | during the study
  Infections
Adverse events related to steroid or cyclophosphamide | during the study
  Adverse events related to steroid or cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Eric THERVET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE, Paris, France

REFERENCES:
- [Result] Pillebout E, Thervet E, Hill G, Alberti C, Vanhille P, Nochy D. Henoch-Schonlein Purpura in adults: outcome and prognostic factors. J Am Soc Nephrol. 2002 May;13(5):1271-8. doi: 10.1097/01.asn.0000013883.99976.22. PMID 11961015
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224
- [Derived] Pillebout E, Alberti C, Guillevin L, Ouslimani A, Thervet E; CESAR study group. Addition of cyclophosphamide to steroids provides no benefit compared with steroids alone in treating adult patients with severe Henoch Schonlein Purpura. Kidney Int. 2010 Sep;78(5):495-502. doi: 10.1038/ki.2010.150. Epub 2010 May 26. PMID 20505654